CLINICAL TRIAL: NCT04621669
Title: A Multi-center, Open-lable, Fixed-sequence Phase I Drug-drug Interaction Clinical Study to Investigate the Pharmacokinetics of SHR3680 With Pgoxin (P-gp Substrates), Rosuvastatin Calcium (BCRP and OATP1B1/1B3 Substrates) and Metformin Hydrochloride (MATE1/2-K Substrates) in Prostate Cancer Patients
Brief Title: Drug-durg Interaction of SHR3680 With Digoxin, Rosuvastatin Calcium and Metformin Hydrochloride
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR3680-I-DDI-03
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Drug-drug Interaction,SHR3680
MeSH Terms: interventions — Digoxin; Rosuvastatin Calcium; Metformin

STUDY DESIGN:
Intervention Model Description: To observe the effect of SHR3680 on the pharmacokinetics of digoxin, Rosuvastatin calcium, metformin hydrochloride and to evaluate the safety. The subjects will take digoxin, Rosuvastatin calcium, metformin hydrochloride at first single dose, then wash out ,and take it at second time together with SHR3680 after multiple administration of SHR3680
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digoxin, Rosuvastatin calcium,SHR3680 (Experimental)
  Interventions: Drug: SHR3680; Drug: digoxin; Drug: Rosuvastatin calcium
- metformin hydrochloride ,SHR3680 (Experimental)
  Interventions: Drug: SHR3680; Drug: metformin hydrochloride

INTERVENTIONS:
Drug: SHR3680 — 240 mg
Drug: digoxin — 0.25 mg
  Arms: digoxin, Rosuvastatin calcium,SHR3680
Drug: Rosuvastatin calcium — 10 mg
  Arms: digoxin, Rosuvastatin calcium,SHR3680
Drug: metformin hydrochloride — 500 mg
  Arms: metformin hydrochloride ,SHR3680

SUMMARY:
The DDI study had been designed to investigate the effect of SHR3680 on the pharmacokinetics of digoxin, Rosuvastatin calcium and metformin hydrochloride

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to enter the study:

1. 18 ≤ age ≤75, male;
2. ECOG score of physical condition is 0 ~ 1;
3. The expected survival time is at least 3 months;
4. Prostate adenocarcinoma confirmed by histological or cytological examination (can be included in mHSPC and mCRPC populations), with no neuroendocrine or small-cell characteristics;CRPC should also meet the following two conditions :(1) serum testosterone level of castration (< 1.7 nmol/L);(2) biochemical progression: prostate-specific antigen (PSA) was increased for 3 consecutive times at an interval of 1 week or more, and increased by more than 50% compared with the lowest value for 2 consecutive times, with PSA > 2 g/L.Or imaging progress: 2 or more new lesions or soft tissue lesions conforming to solid tumor response evaluation criteria were found on bone scan;
5. The functional level of organs must meet the following requirements (no blood transfusion or hematopoietic growth factor treatment was received within 2 weeks before routine blood screening) :

   * the ANC ≧ 1.5 x 109 / L;
   * PLT ≧ 80 x 109 / L;
   * Hb ≧ 90 g/L; 1.5 x ULN - TBIL ≦;
   * ALT and AST≦2.5×ULN;
   * 1.5 x ULN Cr ≦;
   * GFR ≧ 60 ml/min / 1.73 m2.
6. According to the researcher's judgment, it can comply with the experimental scheme;
7. In addition, in accordance with the requirements of regulatory authorities, research centers and relevant departments, and based on the judgment of researchers, you shall be tested for COVID-19 screening when necessary;
8. Volunteer to participate in this clinical trial, understand the study procedures and have signed informed consent.

Exclusion Criteria:

ubjects who meet any of the following criteria will not be admitted to the study:

1. Any previous anti-tumor therapy (including radiotherapy, chemotherapy, surgery, molecular targeted therapy, immunotherapy, etc.), except ADT therapy, shall be completed until the washout period of the first drug administration in this study is <4 weeks;
2. Plan to receive any other anti-tumor therapy during the study;
3. As subjects, to participate in other drug clinical trials, the last trial drug administration is less than 4 weeks from the first administration of the drug in this study (except for the patients who have participated in ADT treatment before and have been out of the group, and the subjects who are still giving free ADT treatment);
4. The presence of intracerebral tumor lesions according to imaging diagnosis;
5. Have a history of epilepsy, or have diseases that can induce epileptic seizures within 12 months before the first administration of the drug in this study (including a history of transient ischemic attack, cerebral stroke (except cerebral ischemia lesions found by simple imaging examination), and need to be hospitalized with cerebral trauma and consciousness disorder);
6. Active heart disease, including severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, and drug-requiring ventricular arrhythmias, within 6 months prior to the first administration of the drug in this study;
7. Inability to swallow, chronic diarrhea and ileus, history of gastrointestinal surgery, or other factors affecting drug use and absorption as determined by the investigator;
8. Patients with active HBV or HCV infection (HBsAg positive and virus copy number ≥500 IU/mL, HCV antibody positive and HCV RNA higher than the lower limit of analytical method detection) and active syphilis;
9. A history of immunodeficiency (including HIV positive, other acquired or congenital immunodeficiency diseases) or a history of organ transplantation;
10. Patients who were unwilling to use effective contraceptive methods during the whole study treatment period and within 3 months after the last administration;
11. Allergic constitution, including a history of severe drug allergy or drug allergy;
12. Screening for excessive smoking in the first 6 months (≥5 cigarettes/day) or smoking within 48 hours before the first dose, or not interrupting smokers during the main study trial, and screening for drug use in the first 3 months with a history of drug abuse or positive drug abuse screening;
13. has a history of alcoholism or within 6 months prior to screening often drinkers, namely the essence of drinking more than 14 units of alcohol a week (1 = 285 mL of alcohol content of 5% beer or 25 mL of 40% alcohol liquor or 100 mL wine alcohol content of 12%) or within 48 h before taking the medicine for the first time drinking, or D - 1 in the alcohol breath test positive, or the body can't stop alcohol intake during the study period;
14. Use of any vitamin product, health product or herb 14 days prior to the first administration;
15. Ingestion of grapefruit or fruit juice products such as grapefruit, foods or beverages containing caffeine, xanthine or alcohol within 48 hours before taking the study drug;Strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, and excretion;
16. Within 2 weeks before the first drug uptake, uptake transporter P-GP, BCRP, OATP1B1/1B3 or MATE1/2-K inhibitors were used, or drugs affecting gastric acid secretion.(Annex I);
17. abnormal coagulation function at screening stage (INR >1.5 or prothrombin time (PT) > ULN+4 seconds or APTT> 1.5uln), bleeding tendency or thrombolytic therapy;
18. Patients with a history of fainting needle or blood, have difficulty in blood collection or cannot tolerate vein puncture for blood collection;
19. Concomitant diseases (such as poorly controlled hypertension, severe diabetes, thyroid disease, psychosis, etc.) or any other conditions that, in the investigator's judgment, would seriously endanger the patient's safety or affect the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-11-19 (Estimated); Primary Completion 2021-05-12 (Estimated); Study Completion 2021-07-05 (Estimated)

PRIMARY OUTCOMES:
Summary of Pharmacokinetic parameters Maximum Plasma concentration (Cmax) for digoxin, Rosuvastatin calcium, metformin hydrochloride | For digoxin and Rosuvastatin calcium group：Day1 and Day22；For metformin hydrochloride group：Day1 and Day19
Summary of Pharmacokinetic parameters Area Under the Plasma Concentration-time Curve form 0 to any time before the last quantifiable concentration(AUC0-t)for digoxin, Rosuvastatin calcium, metformin hydrochloride | For digoxin and Rosuvastatin calcium group：Day1 and Day22；For metformin hydrochloride group：Day1 and Day19
Summary of Pharmacokinetic parameters Area Under the Plasma Concentration-time Curve form 0 to infinite time(AUCinf)for digoxin, Rosuvastatin calcium, metformin hydrochloride | For digoxin and Rosuvastatin calcium group：Day1 and Day22；For metformin hydrochloride group：Day1 and Day19

SECONDARY OUTCOMES:
Tmax of digoxin, Rosuvastatin calcium, metformin hydrochloride | For digoxin and Rosuvastatin calcium group：Day1 and Day22；For metformin hydrochloride group：Day1 and Day19
incidence of adverse events/serious adverse event | From ICF signing date to approximate 2 months
  safety evaluation based on NCI-CTC AE 5.0
T1/2 of digoxin, Rosuvastatin calcium, metformin hydrochloride | For digoxin and Rosuvastatin calcium group：Day1 and Day22；For metformin hydrochloride group：Day1 and Day19
CL/F of digoxin, Rosuvastatin calcium, metformin hydrochloride | For digoxin and Rosuvastatin calcium group：Day1 and Day22；For metformin hydrochloride group：Day1 and Day19
Vz/F of digoxin, Rosuvastatin calcium, metformin hydrochloride | For digoxin and Rosuvastatin calcium group：Day1 and Day22；For metformin hydrochloride group：Day1 and Day19

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qingdao University, Qingdao, China